CLINICAL TRIAL: NCT03073252
Title: The Acute Effect of Egg-Based High Protein Meal on Hypertensive Response to Exercise
Acronym: S47
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Principal Investigator, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 1607017949
Record Dates: First submitted 2017-02-14; First posted 2017-03-08 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Blood Pressure; Cardiovascular Risk Factor

STUDY DESIGN:
Intervention Model Description: subject will consume either the 13g or 30g protein breakfast in a randomized cross-over manner
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Care provider will randomize participants and keep the participant, investigator and outcomes assessor blinded to the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Protein (Experimental): Consumption of normal protein (NP) meal
  Interventions: Other: Normal Protein; Other: HIgh Protein
- High Protein (Experimental): Consumption of high protein (HP) meal
  Interventions: Other: Normal Protein; Other: HIgh Protein

INTERVENTIONS:
Other: Normal Protein — Consumption of a normal protein (NP), egg-based (13 g protein; whole eggs) breakfast bowl
Other: HIgh Protein — Consumption of a high protein (HP), egg-based (30 g protein; whole eggs) breakfast bowl

SUMMARY:
The primary purpose of this study is to explore the effect of high versus normal egg-based protein meals on acute exercise-induced elevated blood pressure.

DETAILED DESCRIPTION:
This study is designed to assess BP changes during and post- exercise after consumption of a test breakfast. The design consists of three visits. The first visit will assess each participants aerobic exercise capacity (VO2 max). Visit 2 and 3 will be clinical testing days where the subject will consume either the 13g or 30g protein breakfast in a randomized cross-over manner and perform the exercise intervention. BP changes will be monitored before and after breakfast consumption, during the exercise intervention,

ELIGIBILITY:
Inclusion Criteria:

* Pre-hypertensive (systolic, 120-139 mm Hg; diastolic, 80-89 mm Hg
* Age ≥ 21
* Body weight <300 lb (136 kg)
* BMI between 20 and 34.9 kg/m2
* Fasting plasma glucose <6.1 mmol/L,
* total cholesterol <6.7 mmol/L
* LDL cholesterol <4.1 mmol/L
* TG <4.5 mmol/L
* No pre-existing or history of cardiovascular, renal or liver disease
* Not currently or previously (past 6 mo) consuming a weight-loss diet or other special/non-balanced diets
* No weight loss/gain (±4.5 kg) within the past 6 mo
* No physical impairments preventing properly exercise execution
* No caffeine intake the day of testing

Exclusion Criteria:

* Hypertensive
* Body weight ≥ 300 lb
* BMI <20 or >35 kg/m2
* Pregnant or planning pregnancy
* Unwilling to consume study foods and beverages
* Fasting plasma glucose ≥6.1 mmol/L
* Total cholesterol ≥6.7 mmol/L
* LDL cholesterol ≥4.1 mmol/L
* TG ≥4.5 mmol/L
* acute illness
* smoking
* diabetic
* pre-existing or history of cardiovascular, renal or liver disease
* currently or previously (past 6 mo) consuming a weight-loss diet or other special/non-balanced diets
* weight loss/gain (±4.5 kg) within the past 6 months
* physical impairments preventing properly exercise execution
* caffeine the day of testing

Ages: 21 Years to 121 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Changes | 6hr testing
  Changes from Baseline to Post Systolic Blood Pressure during 30 minute exercise session

SECONDARY OUTCOMES:
Vasoactive Molecules | 6 hrs
  Vasoactive Molecules analysis using plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
no plans to share data with other researchers